CLINICAL TRIAL: NCT06650969
Title: China Diabetes Cognitive Dysfunction Early Diagnosis and Intervention Study (China-DECODE Study)
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yan Bi, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: DECODE2024
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes; Subjective Cognitive Decline; Mild Cognitive Impairment; Dementia; Cognitive Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction; Dementia | interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — DNA and mRNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Naturalistic observation — Naturalistic observation

SUMMARY:
Type 2 diabetes (T2D) and dementia are both diseases with increasing incidence and prevalence globally, leading to substantial economic burdens for families and society. Notably, diabetes significantly increases the risk of cognitive dysfunction, which is classified into preclinical stage, mild cognitive impairment and dementia based on the disease severity. Cognitive dysfunction is a critical contributor to disability and mortality in elderly diabetes patients. Early diagnosis and intervention are crucial for delaying disease progression, enhancing treatment efficacy, and mitigating the impact of dementia. Currently, research and clinical management of cognitive dysfunction in individuals with diabetes are in their infancy, characterized by limitations such as single-center studies, limited sample sizes, inconsistent diagnostic criteria, and insufficient data sharing. Consequently, clinical diagnosis and treatment strategies are underdeveloped, medical staff's related knowledge is lacking, and potential therapeutic targets remain unexplored. In view of these problems and shortcomings, the population cohort study is supposed to be carried out based on accurate diagnosis and constructed the high standard information and sample bank. The study will establish the standard and quality system of T2D with cognitive dysfunction cohort study (unified standards and norms). The study will integrate the standard biological samples stratified acquisition function module (homogeneity and precision) of cognitive dysfunction in T2D, and complete the construction of biological samples bank and clinical diagnosis and treatment information database. The study will apply and develop brain structural and functional imaging technology to support precision diagnosis of cognitive dysfunction in T2D.

DETAILED DESCRIPTION:
The neuropsychological test battery are used to access the cognitive function of subjects in the study. The laboratory examinations, brain MRI and olfactory function measurements will be done in the screening period. The samples such as plasma, serum, urine and faeces et al. of the subjects will be collected in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years;
* Type 2 diabetes diagnosed according to the American Diabetes Association criteria;
* Willingness and ability to complete systematic neuropsychological tests;
* Understanding of the research procedures and methods, potential benefits and risks of the trial, and sign written informed consent.

Exclusion Criteria:

* Fewer than 6 years of education;
* Left-handedness;
* Dementia;
* Acute metabolic complications such as diabetic ketoacidosis, hyperglycaemic hyperosmolar state and hypoglycaemic coma within the previous 3 months;
* History or presence of neurological or psychiatric disorders;
* Presence of hypothyroidism;
* History of malignancy, or severe kidney or liver dysfunction.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a dynamic prospective cohort study.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2034-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence, incidence of cognitive dysfunction in type 2 diabetes | From 2016 to 2034
  Prevalence, incidence of mild cognitive impairment in type 2 diabetes
Risk factors for cognitive dysfunction in type 2 diabetes, such as diabetes duration, poor glycemic control, hypertension, obesity, dyslipidemia, and active inflammation, et al. | From 2016 to 2034
  Risk factors for the occurrence and progression of mild cognitive impairment in type 2 diabetes, such as diabetes duration, poor glycemic control, hypertension, obesity, dyslipidemia, and active inflammation, et al.
Biomarkers of cognitive dysfunction in type 2 diabetes | From 2016 to 2034
  Diagnostic biomarkers, predictive biomarkers, and prognostic biomarkers of cognitive dysfunction in type 2 diabetes
Glycemic control targets for cognitive dysfunction in type 2 diabetes | From 2016 to 2034
  Glycemic control targets (including glycated hemoglobin, glycemic fluctuations and hypoglycemic events) for slowing or reversing disease progression of cognitive dysfunction in type 2 diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, M.D., Ph.D., Study Director — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (1):
- Department of Endocrinology, Endocrine and Metabolic Disease Medical Center, Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No